CLINICAL TRIAL: NCT01101919
Title: An Open Label, Single And Multiple Dose Study To Investigate The Pharmacokinetics, Safety And Tolerability Of CP-690,550 In Healthy Chinese Subjects
Brief Title: CP-690,550 Pharmacokinetics In Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3921065
Record Dates: First submitted 2010-04-06; First posted 2010-04-12 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-690,550 Dose Group (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Days 1 and 6 dose of 10 mg once daily Days 2-5 doses of 10 mg twice daily

SUMMARY:
This study is designed to evaluate the levels of CP-690,550 in the blood of healthy Chinese subjects following both single doses and multiple doses of drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese Volunteers
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Exclusion Criteria:

* Clinically significant infections within the past 3 months
* Positive screening test for hepatitis B surface antigen, anti-hepatitis C antibody, or human immunodeficiency virus
* Pregnant or nursing women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Single-dose: Cmax, Tmax, t½, AUCinf and AUClast | 1 day
Multiple-dose: Cmin, Cmax, Ctrough, Tmax, t½, AUCtau, and Rac | 5 days

SECONDARY OUTCOMES:
Number of adverse events and number of participants with adverse events | 6 days
Changes in complete blood count and serum chemistry profile | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Beijing, China

REFERENCES:
- [Derived] Krishnaswami S, Wang T, Yuan Y, Alvey CW, Checchio T, Peterson M, Shi H, Riese R. Single- and multiple-dose pharmacokinetics of tofacitinib in healthy Chinese volunteers. Clin Pharmacol Drug Dev. 2015 Sep;4(5):395-9. doi: 10.1002/cpdd.202. Epub 2015 Jul 16. PMID 27137149
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921065&StudyName=CP-690%2C550%20Pharmacokinetics%20In%20Healthy%20Chinese%20Subjects